CLINICAL TRIAL: NCT03775486
Title: A Phase II Randomized, Multi-Center, Double-Blind, Global Study to Determine the Efficacy and Safety of Durvalumab Plus Olaparib Combination Therapy Compared With Durvalumab Monotherapy as Maintenance Therapy in Patients Whose Disease Has Not Progressed Following Standard of Care Platinum-Based Chemotherapy With Durvalumab in First Line Stage IV Non Small Cell Lung Cancer (ORION)
Brief Title: Study of Durvalumab+Olaparib or Durvalumab After Treatment With Durvalumab and Chemotherapy in Patients With Lung Cancer (ORION)
Acronym: ORION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9102C00001; 2018-003460-30 (EudraCT Number)
Record Dates: First submitted 2018-11-27; First posted 2018-12-14 (Actual); Results first posted 2022-12-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer NSCLC
Keywords: NSCLC; Durvalumab; Olaparib; Maintenance; Homologous Recombination Repair (HRR)
MeSH Terms: interventions — durvalumab; olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab/Olaparib Combination Therapy (Experimental): Durvalumab/Olaparib Combination Therapy:
  Durvalumab/SoC chemotherapy (initial therapy phase) followed by Durvalumab/Olaparib (maintenance phase)
  Interventions: Drug: Durvalumab; Drug: Olaparib; Drug: Nab-paclitaxel+carboplatin; Drug: Gemcitabine+carboplatin; Drug: Pemetrexed+carboplatin; Drug: Gemcitabine+cisplatin; Drug: Pemetrexed+cisplatin
- Durvalumab Monotherapy (Experimental): Durvalumab Monotherapy: Durvalumab/SoC chemotherapy (initial therapy phase) followed by Durvalumab/placebo (maintenance phase)
  Interventions: Drug: Durvalumab; Drug: Placebo for Olaparib; Drug: Nab-paclitaxel+carboplatin; Drug: Gemcitabine+carboplatin; Drug: Pemetrexed+carboplatin; Drug: Gemcitabine+cisplatin; Drug: Pemetrexed+cisplatin

INTERVENTIONS:
Drug: Durvalumab — Initial therapy phase: IV infusion q3w for 4 cycles. Maintenance phase: IV infusion q4w.
  Other Names: MEDI4736 (Durvalumab)
Drug: Placebo for Olaparib — Matching tablet
  Other Names: Placebo
  Arms: Durvalumab Monotherapy
Drug: Olaparib — 150-mg tablets (2 × 150-mg tablets for 300-mg dose) 100-mg tablet available if dose reductions are required
  Other Names: AZD2281 (Olaparib)
  Arms: Durvalumab/Olaparib Combination Therapy
Drug: Nab-paclitaxel+carboplatin — Standard of Care chemotherapy (squamous and non-squamous patients)
Drug: Gemcitabine+carboplatin — Standard of Care chemotherapy (squamous patients only)
Drug: Pemetrexed+carboplatin — Standard of Care chemotherapy (non-squamous patients only)
Drug: Gemcitabine+cisplatin — Standard of Care chemotherapy (squamous patients only)
Drug: Pemetrexed+cisplatin — Standard of Care chemotherapy (non-squamous patients only)

SUMMARY:
This is a randomized, double-blind, multi-center, global Phase II study to determine the efficacy and safety of Durvalumab plus Olaparib combination therapy compared with Durvalumab monotherapy as maintenance therapy in patients whose disease has not progressed following Standard of Care (SoC) platinum-based chemotherapy with Durvalumab as first-line treatment in patients with Stage IV non small-cell lung cancer (NSCLC) with tumors that lack activating epidermal growth factor receptor (EGFR) mutations and anaplastic lymphoma kinase (ALK) fusions.

DETAILED DESCRIPTION:
Adult patients with a histologically or cytologically documented advanced NSCLC not amenable to curative surgery or radiation with tumors that lack activation EGFR mutations and ALK fusions are eligible for enrollment. During the initial therapy phase, patients will receive treatment with Durvalumab along with the Investigator's choice of platinum-based doublet therapy for squamous NSCLC (nab-paclitaxel plus carboplatin or gemcitabine plus carboplatin/cisplatin) and non-squamous NSCLC (nab-paclitaxel plus carboplatin or pemetrexed plus carboplatin/cisplatin) for 4 cycles. Patients who have completed 4 cycles and not progressed throughout the initial therapy phase will be randomized in a 1:1 ratio into the maintenance phase of the study to receive either Durvalumab plus placebo or Durvalumab plus Olaparib maintenance therapy. Patients will receive maintenance treatment until specific discontinuation criteria are met, including clinical disease progression (as assessed by the Investigator) or RECIST 1.1-defined radiological Progressive Disease (PD), unacceptable toxicity, and withdrawal of consent. Tumor evaluation scans will be performed until objective disease progression as efficacy assessments. All patients will be followed for survival until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

- Histologically or cytologically documented Stage IV NSCLC not amenable to curative surgery or radiation.

Patients must have tumors that lack activating EGFR mutations and ALK fusions.

* (WHO)/(ECOG) performance status of 0 or 1
* No prior chemotherapy or any other systemic therapy for Stage IV NSCLC
* Adequate organ and marrow function without blood transfusions in the past 28 days,
* At least 1 tumor lesion, not previously irradiated, that can be accurately measured as per RECIST 1.1.

Key Inclusion criteria for randomization to maintenance treatment:

* Documented radiographic evidence of CR, PR, or Stable Disease (SD) as per Investigator-assessed RECIST 1.1 following 4 cycles of platinum-based chemotherapy.
* Creatinine Clearance (CrCl) ≥51 mL/min calculated by the investigator or designee using the Cockcroft-Gault equation or measured by 24-hour urine collection.
* Ability to swallow whole oral medications.
* All patients must provide a formalin-fixed, paraffin embedded tumor sample for tissue-based immunohistochemistry staining and DNA sequencing to determine PD-L1 expression, HRRm status, and other correlatives: either newly acquired or archival tumor samples (<3 years old) are acceptable. If available, a newly acquired tumor biopsy, collected as part of routine clinical practice, is preferred. If not available, an archival sample taken <3 years prior to screening is acceptable. If both an archival sample and a fresh tumor biopsy sample are available, both samples should be submitted for analysis and must be submitted as different samples using different accession numbers. Slides from different blocks cannot be mixed and submitted with the same kit.

Exclusion criteria

* Mixed small-cell lung cancer and sarcomatoid variant NSCLC histology.
* Prior exposure to any chemotherapy agents (except chemotherapy or chemoradiation for non-metastatic disease), polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerase (PARP) therapy, or immunomediated therapy
* Active or prior documented autoimmune or inflammatory disorders.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of Investigational Product (IP)
* untreated (CNS) metastases and/or carcinomatous meningitis
* Active infection.

Exclusion criteria to be randomized to maintenance treatment:

• Inability to complete 4 cycles of platinum-based chemotherapy for any reason or discontinuation of Durvalumab during initial therapy.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2026-09-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, MD, Principal Investigator — Sungkyunkwan University School of Medicine, 135-710, Seoul, Korea
Locations (64):
- United States (9):
  - Research Site, Bonita Springs, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Kansas City, Missouri
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Belgium (3):
  - Research Site, Aalst
  - Research Site, Leuven
  - Research Site, Roeselare
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Farkasgyepü
  - Research Site, Törökbálint
- India (7):
  - Research Site, Ahmedabad
  - Research Site, Jamnagar
  - Research Site, Kochi
  - Research Site, Mysuru
  - Research Site, Nashik
  - Research Site, Pune
  - Research Site, Thiruvananthapuram
- Japan (8):
  - Research Site, Chūōku
  - Research Site, Kanazawa
  - Research Site, Kurume-shi,
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Ube-shi
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Culiacán
  - Research Site, San Luis Potosí City
- Netherlands (3):
  - Research Site, Blaricum
  - Research Site, Harderwijk
  - Research Site, Tilburg
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Prabuty
- Russia (9):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Nal'chik
  - Research Site, P. Herzen Moscow Oncology Rese
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Yaroslavl
- South Korea (5):
  - Research Site, Dongjakgu
  - Research Site, Goyang-si
  - Research Site, Seodaemun-gu
  - Research Site, Seoul
  - Research Site, Suweonsi Paldalgu
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Kharkiv Region
  - Research Site, Kirovohrad
  - Research Site, Odesa
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhia
- United Kingdom (2):
  - Research Site, Dundee
  - Research Site, Hull

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ahn MJ, Bondarenko I, Kalinka E, Cho BC, Sugawara S, Galffy G, Shim BY, Kislov N, Nagarkar R, Demedts I, Gans SJM, Mendoza Oliva D, Stewart R, Lai Z, Mann H, Shi X, Hussein M. Durvalumab in Combination With Olaparib Versus Durvalumab Alone as Maintenance Therapy in Metastatic NSCLC: The Phase 2 ORION Study. J Thorac Oncol. 2023 Nov;18(11):1594-1606. doi: 10.1016/j.jtho.2023.06.013. Epub 2023 Jun 29. PMID 37390980
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9102C00001&attachmentIdentifier=7fc7ec56-03b5-4150-b2a0-175391e8a8e5&fileName=d9102c00001-protocol-redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9102C00001&attachmentIdentifier=22ea3b89-1cbe-40a5-8901-06e2cc9b0847&fileName=d9102c00001-sap-redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9102C00001&attachmentIdentifier=4ac3bc35-f8da-4837-9436-b2bc09aca172&fileName=d9102c00001-study-synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initial therapy phase included participants who received durvalumab in combination with platinum based doublet chemotherapy.
Groups:
- Durvalumab/Olaparib Combination Therapy: Initial Therapy Phase (up to 4 cycles):
  Durvalumab 50 mg/mL intravenous (IV) at a dose of 1500 mg every 3 weeks, and Standard of Care chemotherapy as follows:
  * Nab-paclitaxel: 100 mg/m2 IV on Days 1, 8, and 15 of each 3-week cycle
  * Carboplatin: Area under the concentration-time curve (AUC) 5 or 6 on Day 1 of each 3-week cycle
  * Cisplatin: 75 mg/m2 IV on Day 1 of each 3-week cycle
  * Gemcitabine: 1000 or 1250 mg/m2 IV on Days 1 and 8 of each 3-week cycle
  * Pemetrexed: 500 mg/m2 IV on Day 1 of each 3-week cycle
  Followed by Maintenance Phase:
  Durvalumab 50 mg/mL IV at a dose of 1500 mg every 4 weeks/Olaparib 2 × 150-mg tablets for 300-mg dose twice daily
- Durvalumab/Placebo Therapy: Initial Therapy Phase (up to 4 cycles):
  Durvalumab 50 mg/mL intravenous (IV) at a dose of 1500 mg every 3 weeks, and Standard of Care chemotherapy as follows:
  * Nab-paclitaxel: 100 mg/m2 IV on Days 1, 8, and 15 of each 3-week cycle
  * Carboplatin: Area under the concentration-time curve (AUC) 5 or 6 on Day 1 of each 3-week cycle
  * Cisplatin: 75 mg/m2 IV on Day 1 of each 3-week cycle
  * Gemcitabine: 1000 or 1250 mg/m2 IV on Days 1 and 8 of each 3-week cycle
  * Pemetrexed: 500 mg/m2 IV on Day 1 of each 3-week cycle
  Followed by Maintenance Phase:
  Durvalumab 50 mg/mL IV at a dose of 1500 mg every 4 weeks/matching placebo for oral tablet twice daily
Period: Initial Therapy Phase
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Started | 0 (All 401 participants received the same initial therapy prior to randomization. As such, the subjects listed under the placebo arm for this period are representative of all subjects in the initial therapy phase.) | 401 (All 401 participants received the same initial therapy prior to randomization. As such, the subjects listed under the placebo arm for this period are representative of all subjects in the initial therapy phase.)
Completed | 0 | 269
Not Completed | 0 | 132
Not completed — Other reason provided | 0 | 15
Not completed — Condition under investigation worsened | 0 | 67
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 0 | 34
Not completed — Withdrawal by Subject | 0 | 14
Period: Maintenance Phase
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Started | 134 (All participants received the same initial therapy prior to randomization.) | 135 (All participants received the same initial therapy prior to randomization.)
Participants Who Received Durvalumab | 134 | 134
Participants Who Received Olaparib/Placebo | 128 | 128
Participants Who Terminated the Study | 57 | 57
Completed (Participants ongoing study at data cut-off) | 77 | 78
Not Completed | 57 | 57
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Death | 44 | 45

BASELINE CHARACTERISTICS:
Population: The full analysis set for the maintenance phase is presented
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy | Total
Number analyzed (Participants) | 134 | 135 | 269
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at screening
  Years
    Mean age (years) | 65.9 (9.59) | 63.0 (9.50) | 64.5 (9.64)
Age, Customized [Number; unit: participants] — Age at screening
  participants
    Less than 50 years | 7 | 14 | 21
    Equal to or greater than 50 years to less than 65 years | 49 | 55 | 104
    Equal to or greater than 65 years to less than 75 years | 54 | 54 | 108
    Equal to or greater than 75 years | 24 | 12 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 98 | 97 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 132 | 132 | 264
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 45 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 96 | 89 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking Status [Count of Participants; unit: Participants] — Smoking status at screening
  Participants
    Current | 35 | 31 | 66
    Former | 74 | 72 | 146
    Never | 25 | 32 | 57
Histology Type [Number; unit: participants] — Histology type at screening
  participants
    Squamous Cell Carcinoma | 58 | 59 | 117
    Nonsquamous Cell Carcinoma | 76 | 76 | 152
World Health Organization/Eastern Cooperative Oncology Group [Number; unit: participants] — World Health Organization/Eastern Cooperative Oncology Group measurements at baseline were collected prior to start of maintenance phase.
  participants
    Normal Activity | 52 | 54 | 106
    Restricted Activity | 81 | 80 | 161
    In Bed Less Than or Equal to 50 percent of the Time | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) based on investigator assessments according to Response Evaluation Criteria in Solid Tumours version 1.1.
  PFS is defined as time from date of randomization until the date of objective radiological disease progression using Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) or death (by any cause in the absence of progression).
Time Frame: From randomization until date of objective radiological disease progression or death, or last evaluable assessment in the absence of progression, up to 18 months
Population: Full analysis set (maintenance phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
Participants
  RECIST progression: Target Lesions | 40 | 63
  RECIST progression: Non Target Lesions | 28 | 30
  RECIST progression: New Lesions | 44 | 39
  Death in the absence of progression | 8 | 9
  Censored subjects: Censored RECIST progression | 0 | 0
  Censored subjects: Censored death | 1 | 0
  Censored subjects: Progression-free at time of analysis | 44 | 34
  Censored subjects: Progression-free prior to lost to follow-up | 0 | 0
  Censored subjects: Progression-free prior to withdrawal of consent | 3 | 2
  Censored subjects: Progression-free prior to discontinuation due to other reason | 0 | 0
  Censored subjects: No post-baseline evaluable tumor assessment | 2 | 2
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; Test type: Other; p = 0.074, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.57 to 1.02]
Statistical Analysis 2: Comparison: Durvalumab/Olaparib Combination Therapy; Median progression-free survival (months); Test type: Other; Median = 7.2, 95% CI 2-sided [5.3 to 7.9]
Statistical Analysis 3: Comparison: Durvalumab/Placebo Therapy; Median progression-free survival (months); Test type: Other; Median = 5.3, 95% CI 2-sided [3.7 to 5.8]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) across the maintenance phase.
  OS is defined as time from date of randomization until the date of death by any cause
Time Frame: From randomization until the date of death due to any cause, up to 18 months.
Population: Full analysis set (maintenance phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
Participants
  Death | 44 | 45
  Censored participants (still in survival at follow up or terminated study prior to death) | 90 | 90
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; Test type: Other; p = 0.604, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.59 to 1.36]
Statistical Analysis 2: Comparison: Durvalumab/Olaparib Combination Therapy; Median overall survival (months); Test type: Other; Median = 17.4, 95% CI 2-sided [lower limit 14.1] (NA = insufficient number of participants with events)
Statistical Analysis 3: Comparison: Durvalumab/Placebo Therapy; Median overall survival (months); Test type: Other; Median overall survival (months) = 11.8, 95% CI 2-sided [lower limit 11.8] (NA = insufficient number of participants with events) — The CI lower limit is included as the estimated value as there was an insufficient number of participants with events to calculate a median value

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) defined as number of participants with complete response (CR) or partial response (PR) after randomization
Time Frame: as for outcome 1
Population: Full analysis set for maintenance phase, participants with measurable disease at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 129 | 131
Participants
  Response | 22 | 18
  No Response | 107 | 113

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) defined as time from the date of first documented response following randomization until the first date of documented progression or death in the absence of disease progression.
  Percentage of participants remaining in response at 3, 6, 9 and 12 months estimated using the Kaplan-Meier method.
Time Frame: From date of first documented response until objective radiological disease progression or death, up to 18 months.
Population: Participants with a response and with measurable disease at baseline from the full analysis set (maintenance phase)
Measure: Number; unit: percent
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 22 | 18
percent
  Percentage of participants remaining in response at 3 months | 90.5 | 85.1
  Percentage of participants remaining in response at 6 months | 79.1 | 65.7
  Percentage of participants remaining in response at 9 months | 69.2 | 65.7
  Percentage of participants remaining in response at 12 months | 69.2 | 65.7
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy; Test type: Other — Median duration of response (months); Median duration of response = 6.5, 95% CI 2-sided [lower limit 6.5] (NA = insufficient number of participants with events) — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 2: Comparison: Durvalumab/Placebo Therapy; Test type: Other — Median duration of response (months); Median duration of response = 3.8, 95% CI 2-sided [lower limit 3.8] (NA = insufficient number of participants with events) — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Progression-free Survival in Homologous Recombination Repair Related Gene Mutation (HRRm) Population
Description: Progression-free survival in homologous recombination repair related gene mutation (HRRm) population defined as time from date of randomization until the date of objective radiological disease progression in HRRm population using Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) or death (by any cause in the absence of progression).
Time Frame: as for outcome 1
Population: Full analysis set (maintenance phase); HRRm subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 5 | 9
Participants
  RECIST progression: Target Lesions | 1 | 5
  RECIST progression: Non Target Lesions | 2 | 2
  RECIST progression: New Lesions | 3 | 3
  Death in the absence of progression | 0 | 0
  Censored subjects: Censored RECIST progression | 0 | 0
  Censored subjects: Censored death | 0 | 0
  Censored subjects: Progression-free at time of analysis | 2 | 2
  Censored subjects: Progression-free prior to lost to follow-up | 0 | 0
  Censored subjects: Progression-free prior to withdrawal of consent | 0 | 0
  Censored subjects: Progression-free prior to discontinuation due to other reason | 0 | 0
  Censored subjects: No post-baseline evaluable tumor assessment | 0 | 0
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; Test type: Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.07 to 2.00]
Statistical Analysis 2: Comparison: Durvalumab/Olaparib Combination Therapy; Median progression-free survival (months); Test type: Other; Median (months) = 3.7, 95% CI 2-sided [lower limit 1.7] (NA = insufficient number of participants with events)
Statistical Analysis 3: Comparison: Durvalumab/Placebo Therapy; Median progression-free survival (months); Test type: Other; Median (months) = 3.7, 95% CI 2-sided [1.2 to 16.6]

6. Secondary Outcome: Concentration of Durvalumab
Description: Concentration (pharmacokinetics) of durvalumab
Time Frame: Assessed from start of initial therapy up to 2 years.
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 134
μg/mL
  Cycle 01 Day 01 (Initial Therapy Phase) Post dose: number analyzed (Participants) | 131 | 129
  Cycle 01 Day 01 (Initial Therapy Phase) Post dose | 417.152 (62.694) | 453.724 (43.258)
  Cycle 02 Day 01 (Initial Therapy Phase) Pre dose: number analyzed (Participants) | 129 | 130
  Cycle 02 Day 01 (Initial Therapy Phase) Pre dose | 76.812 (84.586) | 76.959 (71.104)
  Cycle 04 Day 01 (Initial Therapy Phase) Pre dose: number analyzed (Participants) | 127 | 131
  Cycle 04 Day 01 (Initial Therapy Phase) Pre dose | 155.461 (58.251) | 154.947 (50.102)
  Month 03 (Initial Therapy Phase) Pre dose: number analyzed (Participants) | 0 | 0
  Cycle 01 (Maintenance Phase) Post dose: number analyzed (Participants) | 133 | 126
  Cycle 01 (Maintenance Phase) Post dose | 535.078 (40.119) | 524.306 (56.458)
  Cycle 02 (Maintenance Phase) Pre dose: number analyzed (Participants) | 119 | 113
  Cycle 02 (Maintenance Phase) Pre dose | 159.157 (53.813) | 160.315 (54.409)
  Cycle 05 (Maintenance Phase) Pre dose: number analyzed (Participants) | 78 | 77
  Cycle 05 (Maintenance Phase) Pre dose | 166.644 (54.948) | 147.848 (56.204)
  Cycle 08 (Maintenance Phase) Pre dose: number analyzed (Participants) | 55 | 46
  Cycle 08 (Maintenance Phase) Pre dose | 198.932 (47.024) | 154.057 (54.911)
  Cycle 11 (Maintenance Phase) Pre dose: number analyzed (Participants) | 29 | 28
  Cycle 11 (Maintenance Phase) Pre dose | 210.794 (42.117) | 186.092 (39.823)
  Cycle 14 (Maintenance Phase) Pre dose: number analyzed (Participants) | 17 | 11
  Cycle 14 (Maintenance Phase) Pre dose | 276.612 (50.137) | 182.042 (39.341)
  Cycle 17 (Maintenance Phase) Pre dose: number analyzed (Participants) | 7 | 6
  Cycle 17 (Maintenance Phase) Pre dose | 264.096 (55.519) | 217.137 (92.229)
  Cycle 20 (Maintenance Phase) Pre dose: number analyzed (Participants) | 1 | 1
  Cycle 20 (Maintenance Phase) Pre dose | 528.046 | 112.276
  Month 03 (Maintenance Phase) Pre dose: number analyzed (Participants) | 13 | 25
  Month 03 (Maintenance Phase) Pre dose | 12.289 (450.125) | 12.769 (225.898)

7. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Lung Cancer (LC)13
Description: Disease-related symptoms assessed by change from baseline (for maintenance phase) in EORTC QLQ-LC13. Average adjusted mean over first 11 cycles is presented.
  The EORTC QLQ-LC13 was scored according to the published scoring manual. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales in the EORTC QLQ-LC13. Higher scores on symptom scales represent greater symptom severity.
Time Frame: as for outcome 1
Population: Full analysis set (maintenance phase)
Measure: Mean (Standard Error); unit: change from baseline score
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
change from baseline score
  EORTC QLQ-LC13: Dyspnoea: number analyzed (Participants) | 112 | 98
  EORTC QLQ-LC13: Dyspnoea | -1.27 (1.373) | -0.76 (1.500)
  EORTC QLQ-LC13: Coughing: number analyzed (Participants) | 112 | 98
  EORTC QLQ-LC13: Coughing | -2.14 (1.980) | -3.09 (2.172)
  EORTC QLQ-LC13: Pain in chest: number analyzed (Participants) | 112 | 98
  EORTC QLQ-LC13: Pain in chest | 1.31 (1.410) | 3.57 (1.575)
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; EORTC QLQ-LC13: Dyspnoea Estimated difference in adjusted mean change from baseline; Test type: Other; Estimated difference in adjusted mean = -0.51, 95% CI 2-sided [-4.47 to 3.46]
Statistical Analysis 2: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; EORTC QLQ-LC13: Coughing Estimated difference in adjusted mean change from baseline; Test type: Other; Estimated difference in adjusted mean = 0.95, 95% CI 2-sided [-4.81 to 6.71]
Statistical Analysis 3: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; EORTC QLQ-LC13: Pain in chest Estimated difference in adjusted mean change from baseline; Test type: Other; Estimated difference in adjusted mean = -2.26, 95% CI 2-sided [-6.39 to 1.88]

8. Secondary Outcome: Time to Deterioration in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Lung Cancer (LC)13
Description: Disease-related symptoms assessed by time to deterioration (for maintenance phase) in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Lung Cancer (LC)13.
  Symptom deterioration is defined as an increase in the score from baseline of less than or equal to 10) that is confirmed at a subsequent assessment, or death (by any cause) in the absence of a clinically meaningful symptom deterioration.
  NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
Time Frame: as for outcome 1
Population: Full analysis set (maintenance phase)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
months
  EORTC QLQ-LC13: Dyspnoea: number analyzed (Participants) | 134 | 134
  EORTC QLQ-LC13: Dyspnoea | 10.0 [5.6 to 12.2] | 9.7 [6.9 to 12.0]
  EORTC QLQ-LC13: Coughing: number analyzed (Participants) | 132 | 132
  EORTC QLQ-LC13: Coughing | 11.7 [9.3 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 10.6 [7.7 to 12.6]
  EORTC QLQ-LC13: Haemoptysis | 15.0 [11.7 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 12.6 [10.9 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-LC13: Pain In Chest: number analyzed (Participants) | 133 | 134
  EORTC QLQ-LC13: Pain In Chest | 13.8 [10.8 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 11.5 [9.5 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-LC13: Pain In Arm Or Shoulder: number analyzed (Participants) | 131 | 135
  EORTC QLQ-LC13: Pain In Arm Or Shoulder | 15.0 [10.2 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 9.7 [7.4 to 12.6]
  EORTC QLQ-LC13: Pain In Other Parts: number analyzed (Participants) | 128 | 133
  EORTC QLQ-LC13: Pain In Other Parts | 10.3 [8.8 to 12.2] | 10.6 [8.6 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.

9. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire (QLQ) QLQ-C30
Description: Disease-related symptoms and health-related quality of life (HRQoL) assessed by change from baseline (for maintenance phase) in EORTC QLQ-C30. Average adjusted mean over first 11 cycles is presented.
  The EORTC QLQ-C30 was scored according to the published scoring manual. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales, each of the function scales, and the global health status/QoL scale in the EORTC QLQ-C30. Higher scores on the global health status and function scales indicate better health status/function.
  A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / quality of life (QoL) represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time Frame: Includes all assessments occurring within the first 12 months of randomization or until disease progression, up to 18 months.
Population: Full analysis set (maintenance phase)
Measure: Mean (Standard Error); unit: change from baseline score
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
change from baseline score
  EORTC QLQ-C30: Fatigue: number analyzed (Participants) | 112 | 98
  EORTC QLQ-C30: Fatigue | 0.15 (1.327) | -1.49 (1.456)
  EORTC QLQ-C30: Appetite loss: number analyzed (Participants) | 112 | 98
  EORTC QLQ-C30: Appetite loss | -0.13 (1.613) | -3.35 (1.779)
Statistical Analysis 1: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; EORTC QLQ-C30: Fatigue Estimated difference in adjusted mean change from baseline; Test type: Other; Estimated difference in adjusted mean = 1.64, 95% CI 2-sided [-2.20 to 5.47]
Statistical Analysis 2: Comparison: Durvalumab/Olaparib Combination Therapy vs Durvalumab/Placebo Therapy; EORTC QLQ-C30: Appetite loss Estimated difference in adjusted mean change from baseline; Test type: Other; Estimated difference in adjusted mean = 3.22, 95% CI 2-sided [-1.46 to 7.90]

10. Secondary Outcome: Time to Deterioration in EORTC Quality of Life Questionnaire (QLQ) QLQ-C30
Description: Disease-related symptoms and health-related quality of life (HRQoL) assessed by time to deterioration (for maintenance phase) in EORTC QLQ-C30.
  NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
Time Frame: From randomization until date of first symptom deterioration that is confirmed, up to 18 months.
Population: Full analysis set (maintenance phase)
Measure: Median (95% Confidence Interval); unit: time to deterioration (months)
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 135
time to deterioration (months)
  EORTC QLQ-C30: Fatigue: number analyzed (Participants) | 131 | 135
  EORTC QLQ-C30: Fatigue | 8.8 [5.6 to 10.8] | 10 [8.0 to 12.6]
  EORTC QLQ-C30: Nausea And Vomiting | 12.2 [10.2 to 15.0] | 12.6 [9.7 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-C30: Pain: number analyzed (Participants) | 131 | 133
  EORTC QLQ-C30: Pain | 10.2 [7.4 to 12.2] | 9.7 [6.6 to 12.6]
  EORTC QLQ-C30: Dyspnoea: number analyzed (Participants) | 132 | 133
  EORTC QLQ-C30: Dyspnoea | 12.2 [10.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 11.0 [8.8 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-C30: Insomnia: number analyzed (Participants) | 132 | 133
  EORTC QLQ-C30: Insomnia | 13.8 [10.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 10.6 [8.6 to 12.6]
  EORTC QLQ-C30: Appetite Loss: number analyzed (Participants) | 131 | 134
  EORTC QLQ-C30: Appetite Loss | 11.7 [10.1 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 11.5 [10.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-C30: Constipation: number analyzed (Participants) | 132 | 134
  EORTC QLQ-C30: Constipation | 12.2 [10.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 12.0 [10.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  EORTC QLQ-C30: Diarrhoea: number analyzed (Participants) | 133 | 135
  EORTC QLQ-C30: Diarrhoea | 13.8 [10.2 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 11.5 [9.7 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  Physical Functioning | 12.0 [9.3 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 12.0 [9.0 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  Role Functioning: number analyzed (Participants) | 134 | 133
  Role Functioning | 10.0 [5.6 to 12.2] | 10.6 [8.8 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  Emotional Functioning: number analyzed (Participants) | 133 | 135
  Emotional Functioning | 12.2 [9.3 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 11.0 [8.8 to 12.6]
  Cognitive Functioning | 10.2 [6.9 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events. | 10.6 [8.6 to 12.6]
  Social Functioning: number analyzed (Participants) | 134 | 134
  Social Functioning | 9.3 [7.4 to 12.2] | 10.0 [7.7 to NA] — NA is "not applicable". The upper confidence limit was not calculable because of an insufficient number of participants with events.
  Global Health Status/Quality of Life: number analyzed (Participants) | 134 | 133
  Global Health Status/Quality of Life | 10.2 [6.5 to 12.2] | 9.7 [7.4 to 12.0]

11. Secondary Outcome: Presence of Anti-drug Antibodies (ADAs) for Durvalumab
Description: Presence of anti-drug antibodies (ADAs) for durvalumab, as assessed at 3, 6, 12, 16 and 20 weeks after start of treatment and every 12 weeks thereafter until 3 and 6 months after last dose of durvalumab
Time Frame: Assessed from start of initial therapy up to 2 years.
Population: Anti-drug antibody (ADA) evaluable set
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 132 | 130
Participants
  ADA prevalence (any ADA positive, baseline or post-baseline) | 11 | 9
  ADA incidence (treatment-induced or treatment-boosted) | 5 | 4
  ADA positive post-baseline and positive at baseline | 0 | 1
  ADA positive post-baseline and not detected at baseline (treatment-induced) | 5 | 4
  ADA not detected at post-baseline and positive at baseline | 6 | 4
  Treatment-boosted ADA | 0 | 0
  Persistent positive | 0 | 3
  Transient positive | 5 | 2
  Neutralizing anti-drug antibody positive at any visit | 1 | 1

12. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Number of Participants with Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: as for outcome 1
Population: Safety analysis set.
  One participant randomized to the durvalumab/placebo group did not receive any durvalumab or placebo and was excluded from the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
Number analyzed (Participants) | 134 | 134
Participants | 83 | 54

ADVERSE EVENTS:
Time Frame: From randomization until date of objective radiological disease progression or death, or last evaluable assessment in the absence of progression, up to 18 months.
Description: Adverse events and serious adverse events for the safety analysis set during the Maintenance Phase are presented. Deaths for the full analysis set during the Maintenance Phase are presented. The safety analysis set had 1 fewer participant than the full analysis set as 1 participant randomized did not receive durvalumab or placebo and was therefore not included.
  Frequency Threshold for reporting Other Adverse Events: 5 percent
  0 = <5% of events reported
Groups:
- Initial Therapy Phase: Initial Therapy Phase (up to 4 cycles):
  Durvalumab 50 mg/mL intravenous (IV) at a dose of 1500 mg every 3 weeks, and Standard of Care chemotherapy as follows:
  * Nab-paclitaxel: 100 mg/m2 IV on Days 1, 8, and 15 of each 3-week cycle
  * Carboplatin: Area under the concentration-time curve (AUC) 5 or 6 on Day 1 of each 3-week cycle
  * Cisplatin: 75 mg/m2 IV on Day 1 of each 3-week cycle
  * Gemcitabine: 1000 or 1250 mg/m2 IV on Days 1 and 8 of each 3-week cycle
  * Pemetrexed: 500 mg/m2 IV on Day 1 of each 3-week cycle
Arm/Group | Initial Therapy Phase | Durvalumab/Olaparib Combination Therapy | Durvalumab/Placebo Therapy
All-Cause Mortality (participants affected / at risk) | 89/401 | 44/134 | 45/135
Serious Adverse Events (participants affected / at risk) | 104/401 | 25/134 | 19/134
Other Adverse Events (participants affected / at risk) | 368/401 | 116/134 | 104/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Therapy Phase (N=401) | Durvalumab/Olaparib Combination Therapy (N=134) | Durvalumab/Placebo Therapy (N=134)
Abdominal abscess (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 16 | 3 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 13 | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0
Death (General disorders) | 3 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 1
Influenza B virus test positive (Investigations) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 0 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 2 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Therapy Phase (N=401) | Durvalumab/Olaparib Combination Therapy (N=134) | Durvalumab/Placebo Therapy (N=134)
Anaemia (Blood and lymphatic system disorders) | 188 | 35 | 11
Nausea (Gastrointestinal disorders) | 118 | 19 | 10
Decreased appetite (Metabolism and nutrition disorders) | 1 | 16 | 9
Fatigue (General disorders) | 68 | 15 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 13 | 8
Hypothyroidism (Endocrine disorders) | 11 | 8 | 13
Asthenia (General disorders) | 35 | 8 | 10
Vomiting (Gastrointestinal disorders) | 37 | 15 | 3
Weight decreased (Investigations) | 33 | 12 | 6
Alanine aminotransferase increased (Investigations) | 29 | 6 | 11
Diarrhoea (Gastrointestinal disorders) | 53 | 11 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 10 | 4
Pneumonia (Infections and infestations) | 20 | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 49 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 92 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 60 | 0 | 0
Constipation (Gastrointestinal disorders) | 70 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 31 | 0 | 0
Pyrexia (General disorders) | 22 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 23 | 0 | 0
Neutrophil count decreased (Investigations) | 46 | 0 | 0
Platelet count decreased (Investigations) | 21 | 0 | 0
White blood cell count decreased (Investigations) | 25 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years of completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03775486/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03775486/SAP_001.pdf